CLINICAL TRIAL: NCT02795000
Title: Development a Predictive Nomogram for Primary Ovarian Insufficiency
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2014KT1165
Record Dates: First submitted 2016-03-19; First posted 2016-06-09 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2016-06

CONDITIONS: Primary Ovarian Insufficiency
Keywords: Primary Ovarian Insufficiency; nomogram
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood to be retained
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Primary Ovarian insufficiency group: 1. amenorrhea one year or more than one year
  2. amenorrhea more than 4 months and FSH≥40IU/L
  3. ≤42 years old and AMH≤0.071
- The normal group: 1. normal regular menorrhea
  2. ≤42 years old
  3. normal FSH and AMH level

SUMMARY:
The purpose of this research is to develop a predictive nomogram for primary ovarian insufficiency.

DETAILED DESCRIPTION:
Many researches show primary ovarian insufficiency(POI) etiology is related with gene,immunization,iatrogenic, infection factors and social factors etc. In fact, approximate 70-90% POI have no definite cause, so a lot of patients don't know what will happen when they in occult stage of POI. In this research, researchers will investigate all possible factors in POI patients and normal women and select the valuable risk factor by integrated by statistical method to establish the reasonable predictive model.

This study consists two stages.The fist stage is the model establishment, the second stage is the certificate and evaluate the model.

ELIGIBILITY:
Inclusion Criteria:

* Age18--42
* Definite spontaneous last menstrual period
* Informed consent for participating this research and could answer the questionnaires faithfully.

Exclusion Criteria:

* Congenital gonadal dysgenesis and non organic diseases lead to menstrual disorders.
* Endocrine diseases such Polycystic ovary syndrome, hyperprolactinemia, dysfunctional uterine bleeding, low gonadotropin menstrual disorders and hyperthyreosis
* Reproductive toxicity of drugs used
* Release of chemotherapeutic drugs
* Accept sex hormone medicine in recent 3 months
* Pregnant and lactating women
* With serious heart, liver, kidney and other diseases
* With severe psychiatric disorders

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be recruted from gynaecology department clinic of GuangDong provincial hospital of Chinese Medicine and web advertisement from April 2016 and December 2018.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Draw the Primary Ovarian insufficiency normogram | 1years
  Retrospective Investigation on inclusion criteria populations through multivariate cox proportional hazards regression analysis of independent risk factors can enter the predictive model using R software based on regression coefficient related variables draw the corresponding nomogram (nomogram) .

SECONDARY OUTCOMES:
Verify and evaluate the evaluation of Primary Ovarian insufficiency normogram | 2years
  using the bootstrap method nomogram for internal verification to reduce overfitting bias, the evaluation of the model to predict the risk of premature menopause conformity. In the study population data, select postmenopausal cases, the use of prediction of survival analysis model initial assessment model; select Not menopause an independent risk factor for the population were followed ovarian anti-Mullerian hormone (AMH) decreased the extent of menopause Age as a standard curve prediction, evaluation nomogram model predictive accuracy and clinical value of premature menopause, and finally provide the first Chinese people have the physical characteristics of premature menopause prediction model

CONTACTS AND LOCATIONS:
Overall Officials: hongyan Yang, professor, Study Chair — Guangzhou University of Traditional Chinese Medicine
Locations (1):
- Guangdong provicial hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided